CLINICAL TRIAL: NCT00655694
Title: A Non Interventional Study to Asses the Utility of Genomic/ Proteomic/ Metabonomic Profiling Approaches to the Classification and Pathological Basis of Inflammatory Lung Disease in Smokers, and Ex-smokers vs. Non-smokers and Asthmatics
Brief Title: Genomic/ Proteomic/ Metabonomic Profiling in Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Type: Observational
Why Stopped: Lead Researcher left the Department
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 05/Q0410/97
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; smokers; healthy volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Specimen Collection; Urination; Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: sputum, blood, urine, exhaled breath, lung function

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic disease characterized by progressive airflow obstruction, chronic cough and dyspnoea in advanced stages.

We hope to develop a better understanding of lung disease. Information from these studies will only be used for research purposes, to help develop safer and more effective treatments for asthma and COPD.

DETAILED DESCRIPTION:
Techniques such as genomics, proteomics and metabonomics, Technologies that aim to identify and quantify the dynamic set of all small molecules and metabolites present in an organism or a biological sample, offer the prospect of efficiently distinguishing individuals with particular diseases. The advantages of proteomics and metabonomics is that it can be carried out on a standard preparation of serum, plasma or urine, circumventing the need for specialist preparation of cellular mRNA required for genomics This methodology is based on mass spectrometry (MS), gas chromatography-mass spectrometry (GC-MS), and nuclear magnetic resonance (NMR) to analyze metabolites. High-performance liquid chromatography (HPLC) may also be applied. Several peak alignment algorithms have been developed to match the chromatograms before applying pattern recognition. Based on the pattern recognition, several potential biomarkers may be found and further identified by MS.. Finally, a number of potential biomarkers will be identified for distinguishing asthma and COPD.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria - Healthy non-smokers

  * Non-smoking volunteer aged 40 -75 years (age matched to COPD patients)
  * Normal spirometry (FEV1/FVC ratio >70% and FEV1>80% predicted)
  * Subjects are able to give informed consent Inclusion Criteria-COPD patients (stage 2-3 according to the GOLD guidelines)
  * Current and/or ex-smokers with no less than 10 pack-year smoking history aged 40-75 years
  * 30% FEV1 < 80% of predicted (the upper value is a postbronchodilator value)
  * FEV1/FVC < 70%
  * Stable COPD (no chest infection requiring antibiotics and/ or oral steroids in the past 2 months)
  * Long-acting beta2-agonists and long-acting antimuscarinic bronchodilators need to be stopped at least 8 hours before the study visit
  * The subjects are able to give informed consent
* Inclusion Criteria - healthy smokers

  * Current smokers aged 40 -75 years (age matched to COPD patients)
  * Normal spirometry (normal FEV1/FVC ratio >70% and FEV1>80% predicted)
  * Subjects are able to give informed consent
* Inclusion Criteria - asthmatics

  * Non-smoking asthma patients aged 40 -75 years (age matched to COPD patients)
  * Normal spirometry (normal FEV1/FVC ratio >70% and FEV1>80% predicted)
  * Subjects are able to give informed consent

Exclusion Criteria:

* Exclusion Criteria - Healthy non-smokers

  * Chest infection that required treatment with antibiotics within the last 4 weeks
  * Subjects who have received research medication within the previous one month
  * Subjects unable to give informed consent
  * Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study Exclusion Criteria-COPD patients
  * Bronchodilator reversibility > 12%
  * Chest infection that required treatment with antibiotics within the last 4 weeks
  * Subjects who have received research medication within the previous one month
  * Subjects unable to give informed consent
  * Patients with significant co-morbidities including any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study as judged by the investigator
  * Any other respiratory disease, which is considered by the investigator to be clinically significant
* Exclusion Criteria - healthy smokers

  * Chest infection that required treatment with antibiotics within the last 4 weeks
  * Subjects who have received research medication within the previous one month
  * Subjects unable to give informed consent
* Exclusion Criteria - asthmatics

  * Chest infection that required treatment with antibiotics within the last 4 weeks
  * Patients with significant co-morbidities as judged by the investigator
  * Subjects who have received research medication within the previous one month
  * Subjects unable to give informed consent

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01 (Estimated); Primary Completion 2007-09 (Estimated); Study Completion 2007-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — National Heart and Lung Institute
Locations (1):
- National Heart and Lung Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No